CLINICAL TRIAL: NCT00967265
Title: Introduction Seminar About Patient Participation and Treatment Options for Patients on Waiting List in a Community Mental Health Centre - Development, Effect, Experiences and Costs
Brief Title: Introduction Seminar About Patient Participation and Treatment Options for Psychiatric Patients on Waiting List
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Introduction seminar
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Mental Disorders
Keywords: Introduction seminar; Psychoeducation; Waiting list; Patient participation; Mental disorders
MeSH Terms: conditions — Mental Disorders; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Introduction seminar (Experimental): Psychoeducation for patients on waiting list
  Interventions: Behavioral: Introduction seminar
- Usual care (Active Comparator): Usual care
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Introduction seminar — The seminar will be held over two half days, each lasting 2.5 hours. Up to 30 patients can participate in each seminar. The details of the content of the program will be developed based on study one. The preliminarily plans are to give general information about the community mental health centre, the available treatment options and patients rights by presentations from health personnel and user representatives. At the end of each day, the patients will be divided into small groups mentored by health personnel were they can discuss the presentations and ask questions. In the breaks, literature and other type of information for patients will be on display. All participants will get a folder with details of the program and leaflets from patient organisations and governmental agencies.
  Other Names: psychoeducation
  Arms: Introduction seminar
Other: Usual care — Usual care
  Arms: Usual care

SUMMARY:
Patient participation is a central concept in Norwegian health policy. It is mandatory in hospitals and emphasised as one of the most prioritised areas by the Government. Studies from Norway have repeatedly found that patients who seek help in community mental health centres ("DPS") are dissatisfied with the information they receive and about their possibility for real influence in their treatment.

One way to improve individual patient participation might be to give patients information before they start their treatment. This can be done as group based patient education to reduce the resources needed. Furthermore, as there are waiting lists for treatment, such introduction seminars could be held while patients are waiting to use this time in a meaningful way.

The present study therefore aims at testing the effect of an introduction seminar for patients on waiting list in a community mental health centre.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years referred for out patient treatment who get a guarantee of starting treatment between 2 and 6 months will be included.

Exclusion Criteria:

* patients with a guarantee of starting treatment in less than two months and
* patients who do not understand the consequences of taking part in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-06; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Behavior and symptoms | 12 months
  Behavior and Symptom Identification Scale (BASIS-32)
knowledge on treatment preference | 1 month
patient activation (coping) | 4 months
  measured with Patient Activation Measure (PAM)

SECONDARY OUTCOMES:
Client satisfaction | Baseline, 4 and 12 months
  Satisfaction measured with Client Satisfaction Questionnaire (CSQ-8)
Perceived participation | Baseline, 4 and 12 months
  Perceived participation measured with Perception of care (PoC)
Psychiatric Out-Patient Experiences | Baseline, 4 and 12 months
  Psychiatric Out-Patient Experiences Questionnaire (POPEQ)
Quality of Life | Baseline, 4 and 12 months
  WHO-5
motivation for treatment | Baseline, 1 and 4 months
  motivation for treatment (questions)
costs | Baseline, 1, 4 and 12 months
  data on health care use, sick leave, medication and other direct and indirect costs will be collected
Knowledge | Baseline, 1, 4 and 12 months
  measured using a self developed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Tiller DPS, Trondheim, Norway

REFERENCES:
- [Result] Koksvik JM, Linaker OM, Grawe RW, Bjorngaard JH, Lara-Cabrera ML. The effects of a pretreatment educational group programme on mental health treatment outcomes: a randomized controlled trial. BMC Health Serv Res. 2018 Aug 29;18(1):665. doi: 10.1186/s12913-018-3466-2. PMID 30157839